CLINICAL TRIAL: NCT06304285
Title: A Study Assessing the Effects of Acupuncture in Parkinson's Disease Patients With Chronic Appendicitis: a Single-center, Randomized, Double-blind Study
Brief Title: A Study Assessing the Effects of Acupuncture in Parkinson's Disease Patients With Chronic Appendicitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-ky421
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Disease; Chronic Appendicitis; Acupuncture
Keywords: Parkinson's disease; acupuncture
MeSH Terms: conditions — Parkinson Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): The subjects received acupuncture treatment at the following points: Tianshu, Zusanli, Hegu, Taichong, Shangjuxu, Jigou, Zhaohai, Lanwei and shousanli.
  Interventions: Other: Acupuncture treatment
- control group (Sham Comparator): Treatment with comfort needle and comfort embedding needle
  Interventions: Other: Sham acupuncture treatment

INTERVENTIONS:
Other: Acupuncture treatment — Acupuncture was performed according to the corresponding acupoint of the patient
  Arms: Acupuncture group
Other: Sham acupuncture treatment — The needle only touches the patient's skin and does not penetrate the skin
  Arms: control group

SUMMARY:
The incidence of PD is high, and when the disease is serious to a certain extent, the effect of drugs to control symptoms decreases, resulting in a significant reduction in the quality of life of patients. Recent studies have found that these PD symptoms are closely related to the intestine. For several cases of PD syndrome patients complicated with chronic appendicitis, our research group conducted acupuncture on points related to constipation and chronic appendicitis, and found that constipation and related motor symptoms of patients could be significantly improved. Clinical studies have shown that acupuncture also has a certain therapeutic effect on non-motor symptoms of Parkinson's disease, such as anxiety and depression, decreased olfactory function, sleep disorders, constipation, early skeletal muscle pain, cognitive dysfunction, etc., which can delay the progression of the disease and improve the quality of life of patients. Starting from intestinal acupuncture, this project further clarified the role of acupuncture treatment in the comprehensive treatment of PD

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with bradykinesia, combined with resting tremor and/or myotonia.
* Appendix CT suggested chronic appendicitis evaluated by two experienced experts.
* All subjects and their guardians give informed consent to the content of this study and sign informed consent.
* Normal coagulation function.
* If the patient had taken oral anti-PD drugs, it had been stable for at least 2 weeks at enrollment.

Exclusion Criteria:

* Treatment with dopamine blockers or dopamine depleters in doses and time courses consistent with drug-induced parkinsonism.
* Neuroimaging examination of presynaptic dopaminergic system function was normal.
* Patients who had suffered severe brain trauma or underwent complex craniotomy within 5 years prior to enrollment.
* Cognitive disorders that are not on the Parkinson's spectrum, such as Alzheimer's disease, frontotemporal dementia, and Niemann-Pick disease, have been diagnosed.
* People diagnosed with severe neuropsychiatric disorders (epilepsy, bipolar disorder, major depressive episode, etc.) according to DSM-V.
* Complicated with serious systemic diseases, disorders of consciousness, stroke, serious coronary heart disease, diabetes, liver and kidney diseases, and serious visual and hearing disorders.
* Patients with severe organic or functional dysphagia;Those who were deemed by the researcher to be unable to complete the visit and auxiliary examination as required by the study protocol.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Score of MDS Unified-Parkinson Disease Rating Scale III | 3 month
  The changes of MDS-UPDRS III scores before and after acupuncture treatment were compared.The lowest score was 0 and the highest was 132, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhua Chen, M.M.S., Study Chair — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No